CLINICAL TRIAL: NCT04017442
Title: Neuraxial Preservative Free Morphine for Normal Spontaneous Vaginal Delivery: A Prospective Double Blind Randomized Control Trial
Brief Title: Neuraxial Preservative Free Morphine for Normal Spontaneous Vaginal Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Daniel Katz, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 18-2789
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Postpartum Pain; Postpartum Depression; Opioid Consumption
Keywords: Postpartum depression; Postpartum anxiety; Postpartum opioids
MeSH Terms: conditions — Depression, Postpartum | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind, prospective, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only individual that will know to which group the patient was assigned is the individual on the study team who is drawing up the medication. This individual will have no other role in the assessment or evaluation of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Morphine (Experimental): 2mg preservative free morphine
  Interventions: Drug: Preservative Free Morphine
- Saline (Placebo Comparator): 4 mL preservative free saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Preservative Free Morphine — After delivery of the baby patients will receive via the epidural catheter prior to its removal.
  Arms: Morphine
Drug: Saline — After delivery of the baby patients will receive via the epidural catheter prior to its removal.
  Other Names: Placebo
  Arms: Saline

SUMMARY:
Patients presenting for normal spontaneous vaginal delivery who have a neuraxial anesthestic will be randomized to receive preservative free morphine or saline placebo after delivery.

DETAILED DESCRIPTION:
After obtaining consent, women presenting to the labor floor at Mount Sinai Hospital will be randomized into two groups, intervention and placebo. Baseline demographic data and surveys in regards to postpartum depression, anxiety, breastfeed willingness and pain scores will be obtained. After delivery of the baby patients will either receive 2mg preservative free morphine or saline via the epidural catheter prior to its removal. The study team will then record pain and recovery scores, as well as follow up screens to the aforementioned endpoints. The study will end at the 6 week postpartum visit with the patient's obstetrician.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in labor

Exclusion Criteria:

* Not a candidate for neuraxial anesthesia
* Patient refusal
* Allergy to morphine
* Patients with chronic pain syndromes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Katz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine: 2mg preservative free morphine (4mL) via the epidural catheter within 1 hour of vaginal delivery
- Saline: 4 mL preservative free saline via the epidural catheter within 1 hour of vaginal delivery
Period: Overall Study
Arm/Group | Morphine | Saline
Started | 80 | 80
Completed | 59 | 58
Not Completed | 21 | 22
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Saline | Total
Number analyzed (Participants) | 80 | 77 | 157
Age, Continuous [Median (Full Range); unit: years] | 33.0 [18.0 to 47.0] | 33.0 [21.0 to 51.0] | 33.0 [18.0 to 51.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 77 | 157
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 44 | 40 | 84
  African American | 8 | 7 | 15
  Asian | 9 | 12 | 21
  Hispanic/Latino | 12 | 10 | 22
  Other | 7 | 7 | 14
  Missing | 0 | 1 | 1
BMI [Median (Full Range); unit: kg/m^2] | 29.3 [19.5 to 54.9] | 28.7 [20.5 to 63.6] | 29.1 [19.5 to 63.6]
Weight [Median (Full Range); unit: lbs] | 175 [117 to 300] | 165 [105 to 394] | 170 [105 to 394]
Height [Median (Full Range); unit: inches] | 65.0 [60.0 to 71.0] | 64.0 [59.0 to 71.0] | 64.0 [59.0 to 71.0]
Gestational Age [Median (Full Range); unit: weeks] | 39.4 [35.6 to 41.6] | 39.3 [34.4 to 41.4] | 39.3 [34.4 to 41.6]
Gravidity [Count of Participants; unit: Participants]
  1 | 33 | 28 | 61
  2 | 18 | 18 | 36
  3 | 16 | 10 | 26
  >3 | 13 | 21 | 34
Parity [Count of Participants; unit: Participants]
  0 | 45 | 36 | 81
  1 | 20 | 23 | 43
  2 | 8 | 7 | 15
  3 | 5 | 3 | 8
  >3 | 2 | 8 | 10
The Edinburgh Postnatal Depression Scale (EPDS) [Median (Inter-Quartile Range); unit: units on a scale] — A 10-item instrument to assess postpartum depression, with total score from 0-30. Higher score indicates more depressed symptoms.
  units on a scale | 4 [1 to 6] | 3 [1 to 6] | 3 [1 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption in MME
Description: Quantity of opioid in morphine milligram equivalents (MME) used within 24 hours of delivery.
  The conversions from opioids to MME were as follows: 2 mg oral hydromorphone as 8 MME, 5 mg oxycodone 7.5 MME. To convert the PO hydromorphone to MME, IV hydromorphone was converted to morphine with a 4:1 ratio to convert to morphine followed by a 1:3 ratio to convert IV to PO.
Time Frame: within 24 hours of delivery
Measure: Median (Full Range); unit: MME
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 80 | 77
MME | 0 [0 to 47.5] | 0 [0 to 72]

2. Secondary Outcome: Pain Score
Description: Pain Score: Likert full scale 0-10, with higher score indicating more pain
Time Frame: at 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 75 | 70
score on a scale | 2 [1 to 4] | 3 [1.5 to 5]

3. Secondary Outcome: Obstetric Quality of Recovery Score (OBSQ10)
Description: OBSQ10 total score 0-100, with higher score indicating better health status
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 80 | 77
score on a scale | 77 [60 to 90] | 85 [71 to 92]

4. Secondary Outcome: Number of Participants With Edinburgh Postnatal Depression Scale (EPDS) >10
Description: Number of Participants with positive EPDS screen in the 6-week post-delivery EPDS defined as a score higher than 10.
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item instrument to assess postpartum depression, with total score from 0-30. Higher score indicates more depressed symptoms.
Time Frame: up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 80 | 77
Participants | 7 | 5

5. Secondary Outcome: Number of Participants With Exclusive Breast Feeding
Description: Participants will respond yes/no as to their breast feeding success and continuation exclusively.
Time Frame: 1 week
Population: some participants lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Saline
Number analyzed (Participants) | 80 | 77
Participants
  1 week: number analyzed (Participants) | 75 | 70
  1 week | 22 | 26
  6 weeks: number analyzed (Participants) | 59 | 58
  6 weeks | 26 | 22

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Morphine | Saline
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/77
Other Adverse Events (participants affected / at risk) | 0/80 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04017442/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04017442/ICF_001.pdf